CLINICAL TRIAL: NCT02315378
Title: Anxiety Reduction Treatment for Acute Trauma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The original PI, Alexander Neumeister, left NYULMC. No data was analyzed.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-01334; W81XWH-08-1-0412 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2016-08

CONDITIONS: Anxiety
Keywords: Anxiety, Acute Trauma
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARTAT (Other): A one-session intervention targeting at-risk individuals (those continuing to experience peritraumatic panic following a trauma) and designed to reduce peritraumatic anxiety and enhance self-efficacy.
  Interventions: Behavioral: ARTAT
- TAU (Other): Treatment as Usual
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: TAU — Treatment as Usual for patients presenting after accidents and assaults as it pertains to mental health, is a brief intervention that varies in length depending on the patient's needs. If the patient is highly distressed, the social worked will provide brief crisis management support. The social worker also performs case management functions such as attempting to get in touch with family, contacting shelter or hotel if the patient is homeless, contacting other social service agencies if needed, and providing the patient referrals for mental health services in the community. A psychiatrist will also be called to assess the patient only if he or she appears to be a threat to self (suicidal) or others, and exclusion criteria for this study.
  Other Names: Treatment as Usual
  Arms: TAU
Behavioral: ARTAT — A one-session intervention targeting at-risk individuals (those continuing to experience peritraumatic panic following a trauma) and designed to reduce peritraumatic anxiety and enhance self-efficacy.
  Other Names: Anxiety Reduction Treatment for Acute Trauma
  Arms: ARTAT

SUMMARY:
This study is a randomized controlled trial to investigate the feasibility and effectiveness of a brief Anxiety Reduction Treatment for Acute Trauma (ARTAT) with adults (over age 18) showing signs of peritraumatic anxiety in the Emergency Department of Bellevue Hospital, New York in the hours following a psychologically traumatic event. Thirty-six participants will be enrolled over a 12-month period: 18 receiving ARTAT and 18 receiving Treatment As Usual (TAU). The study will target anxious arousal in patients immediately (1 to 8 hours) following a trauma. Participants will be recruited from among patients who present in the Emergency Department at Bellevue Hospital for treatment of an injury sustained in a traumatic event (accident, assault) as long as injuries do not preclude participation. Participants included in the study will have experienced a trauma within 8 hours and presenting with signs of a strong risk factor for PTSD: peritraumatic panic (severe psychological and physiological anxiety symptoms such as fear of dying, fear of losing emotional control, tachycardia, sweating, shaking and dissociation symptoms such as derealisation and depersonalization that occur during and immediately following a trauma. Following the initial assessment, eligible participants will be randomized to receive the one-hour anxiety-reduction intervention designed to reduce anxiety and panic symptoms through education and anxiety y management skills or TAU. The clinician administered and self-report assessments will be conducted at screening, baseline, post-treatment, weekly, and at a one-month and three-month follow-up.

DETAILED DESCRIPTION:
The purpose of the proposed research is to pilot a behavioral intervention specifically designed to reduce the symptoms of peritraumatic panic, in order to reduce the likelihood of subsequent PTSD. The investigators have developed the Anxiety Reduction Treatment for Acute Trauma (ARTAT), a one-session intervention targeting at-risk individuals (those continuing to experience peritraumatic panic following a trauma) and enhance self-efficacy. The intervention provides education about common responses to trauma in order to normalize symptoms and teaches individuals anxiety management techniques such as deep breathing and muscle relaxation. ARTAT specifically avoids encouraging people to process the trauma (given evidence that this may enhance arousal).

This study is a randomized controlled trial of a single session 60- minute Anxiety Reduction Treatment for Acute Trauma (ARTAT) administered during Emergency Department (ED) admission to patients presenting with anxiety following traumatic exposure. Thirty-six participants will be enrolled over a 12-month period (18 receiving ARTAT and 18 receiving TAU). The study will target anxious arousal in patients immediately (1 to 8 hours) following a trauma. Participants will be recruited from among patients who present in the Bellevue Emergency Department for treatment of an injury sustained in a traumatic event (accident, assault) as long as injuries do not preclude participation. Participants included in the study will have experienced a trauma within 8 hours and presenting with signs of a strong risk factor for PTSD: peritraumatic panic (severe psychological and physiological anxiety symptoms such as fear of dying, fear of losing emotional control, tachycardia, sweating, shaking and dissociation symptoms such as derealisation and depersonalization that occur during and immediately following a trauma. Following the initial assessment, eligible participants will be randomized to receive the one-hour anxiety-reduction intervention designed to reduce anxiety and panic symptoms through education and anxiety y management skills or the TAU. The clinician administered and self-report assessments will be conducted at screening, baseline, post-treatment, and at a one-month and three-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have experienced an acute psychologically traumatic event within the last 8 hours
* Resting hear rate of 80 BPM or greater upon ED presentation

Exclusion Criteria:

* Attending physician does not concur with enrolling subject in study
* Traumatic event occurred more than 8 hours before ED arrival
* Physical injury that contraindicates participation
* Significant head injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Acute Stress Disorder (ASD) Interview | up to one month
  Structured clinical interview that is based on the DSM-IV criteria for acute stress disorder.
Clinician Administered PTSD Scale (CAPS) | up to three-month follow-up
  Structured clinical interview used to determine PTSD diagnosis.
Structured Clinical Interview for DSM-IV | one-month to determine life history of PTSD
  Interview to determine the presence of current or past DSM-IV Axis I disorders.
Event Severity Rating Scale (ESR) | Baseline
  Questionnaire that includes 6 items assessing the intensity of experiences during the event, including extent of injury, life threat to self or loved ones, witnessing injury or death, exposure to horrifying scenes, and an overall how sever the event was.
Mini-Mental status Exam (MMSE) | Screen
  This is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language with a maximum score of 30.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BA1) | Baseline, post-treatment, one-month and three month follow-up
  A 21 item measure that assesses the severity of the subjects anxiety, addressing both the physiological and cognitive components of anxiety
Peritraumatic Dissociative Experiences Questionnaire (PDEQ) | Baseline
  A 10 item measure of dissociative symptoms
Peritraumatic Distress Inventory (PDI) | Baseline
  Assesses respondents' emotional and physical reactions experienced during or immediately after a traumatic event.
Life Stressor Checklist - Revised (LSC-R) | one-month follow-up
  This is a 30-item screening measure of exposure to stressful events across the lifespan, including events such as a physical assault, sexual assault, being robbed or mugged, and the catastrophic death of a loved one.
Posttraumatic Stress Disorder Checklist - Specific Stressor Version (PCL-S) | one-month and three-month follow-ups
  Assesses PTSD symptomatology and severity in response to respondents' traumatic event.

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Marmar, MD, Principal Investigator — NYU School of Medicine